CLINICAL TRIAL: NCT03660761
Title: Efficacy and Safety of Apatinib Combined With Dose-dense Temozolomide in Recurrent Glioblastoma
Brief Title: Apatinib in Recurrent or Refractory Intracranial Central Nervous System Malignant Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rongjie Tao (Other)
Responsible Party: Sponsor-Investigator, Rongjie Tao, Clinical Professor, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShandongCHI005
Record Dates: First submitted 2018-08-11; First posted 2018-09-07 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Efficacy and Safety
MeSH Terms: interventions — apatinib; Temozolomide

STUDY DESIGN:
Intervention Model Description: single arm
Masking Description: Open Label (Subject)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- apatinib 500mg (Experimental)
  Interventions: Drug: apatinib; Drug: temodar

INTERVENTIONS:
Drug: apatinib — The patient was given a daily dose of apatinib 500mg (or based on weight). For adult, the dose of apatinib was prescribed with 425 mg or 500 mg per day and four weeks for a cycle. The dosage was modified to 250 mg if patients experienced ≧grade 2 hematologic adverse events, hand and foot syndrome, proteinuria, fecal ocular blood, or grade 3/4 hypertension, or other grade 3/4 adverse events. Apatinib was administrated until disease progression, unacceptable toxicity or death.
Drug: temodar — dose-dense temozolomide (100 mg/m2 , 7 days on with 7 days off ) , 28d

SUMMARY:
The patient was given a daily dose of apatinib 500mg (or based on weight). Individualized chemotherapy regimens were given based on molecular expression and prior chemotherapy.

DETAILED DESCRIPTION:
The patient was given a daily dose of apatinib 500mg (or based on weight). Individualized chemotherapy regimens were given based on molecular expression and prior chemotherapy. Brain MRI+MRS was examined every 3 months; Blood routine, urine routine and liver and kidney function were examined once a week.

ELIGIBILITY:
Inclusion Criteria:

* (1) 18 years < the age of patients > 70 years. (2) Karnofsky performance scale (KPS) ≥ 60. (2) Histologically confirmed diagnosis of GBM World Health Organization [WHO] Grade IV. (3) They were required to have measurable or evaluable disease by magnetic resonance imaging (MRI) confirmation and a minimum life expectancy of 8 weeks. (4) Definition of relapse: all patients must have progressive disease on MRI defined by Response Assessment in Neuro-Oncology (RANO) criteria after the standard Stupp protocol. The time interval for the start of treatment was at least 12 weeks from prior radiotherapy unless there was either histopathologic confirmation of recurrent tumor or new contrast enhancement on MRI outside of the radiotherapy treatment field. (5) Adequate bone marrow function (leukocyte count ≥ 4000/μL, neutrophil count ≥1500/µL, platelet count ≥100 000/µL, hemoglobin ≥8.0g/dL), adequate renal function (serum creatinine ≤ 150μmol/L, 24 hours urine protein ≤3.4g), and liver function (total bilirubin ≤34μmol/L and aspartate and alanine aminotransferase ≤120U/L).

Exclusion Criteria:

* (1) extracranial metastatic disease, (2) Gliadel wafer treatment, (3) severe cardiopulmonary insufficiency, (4) status epilepticus, (5) pregnancy, (6) gastrointestinal bleeding, (7) uncontrolled blood pressure with medication (>140/90 mm Hg), (8) swallowing difficulties. (9) HIV positivity with a combination antiretroviral therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2018-01-06 (Actual)

PRIMARY OUTCOMES:
Response to treatment | up to 3 months
  Response were evaluatedevery 1-3 months with Response Evaluation Criteria in Solid Tumors version 1.0 (RECIST 1.0) usingdynamic contrast enhancement magnetic resonance imaging (MRI) or computed tomography (CT). Complete response (CR) was defined as complete disappearance of target lesions and maintaining ≥ 4 weeks; partial response (PR): ≥ 30% reduction in maximum diameterof tumor and keepingstable ≥ 4 weeks; progressive disease (PD):>20% increase in bidimensionalmeasurements of the lesions, or emerging one or more newlesions; stable disease (SD): criteria for CR, PR and PDnot met.PFS was defined as the initial treatment to the disease progression or the date of death.

SECONDARY OUTCOMES:
Median non-progress survival (PFS) | up to 12 months
  Median non-progress survival (PFS)

CONTACTS AND LOCATIONS:
Locations (1):
- Neurosurgery, Shandong Cancer Hospital and Institute, Jinan, Shandong, China

REFERENCES:
- [Result] Kasper H. [The supplying of vitamin A after pancreatectomy]. Med Welt. 1968 Jan 20;3:178-80. No abstract available. German. PMID 5728925
- [Result] Potapova TV, Sharovskaia IuIu, Kovalev SA, Mittel'man LA, Chailakhian LM. [Effect of the ion composition of the surrounding medium on membrane potentials of L cells]. Tsitologiia. 1972 Nov;14(11):1335-41. No abstract available. Russian. PMID 4654530